CLINICAL TRIAL: NCT01090076
Title: The Use of Specialised Amino Acid Mixture in Pressure Ulcer Wound Healing Rates-A Placebo Controlled Trial
Brief Title: The Use of Specialised Amino Acid Mixture in Pressure Ulcer Wound Healing Rates- A Placebo Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Alvin Wong, Senior Dietitian, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ABOUND
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer Wound; Specialized Amino Acid Mixture
MeSH Terms: conditions — Pressure Ulcer | interventions — Arginine; Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abound (Experimental): Abound (7 g of Arginine, 7 g Glutamine and 1.2 g HMB)
  Interventions: Dietary Supplement: Abound (7 g of Arginine, 7 g Glutamine and 1.2 g HMB)
- Placebo (Placebo Comparator): Placebo comparator that contains none of the active ingredients
  Interventions: Dietary Supplement: Abound (7 g of Arginine, 7 g Glutamine and 1.2 g HMB)

INTERVENTIONS:
Dietary Supplement: Abound (7 g of Arginine, 7 g Glutamine and 1.2 g HMB) — Active Arm : Abound x 2 sachets/d (Each sachet provides additional 7g L-Arginine, 7g L-Glutamine, 1.2 g HMB and 79 Kcal) Placebo Arm: Abound(placebo) x 2 sachets/d

SUMMARY:
This research aims to address the gap in the studies done and test the effects of a commercial mixture of 7 g of Arginine, 7 g Glutamine and 1.2 g HMB* twice a day on hard to heal pressure ulcers in an Asian patient cohort in an acute healthcare setting.

DETAILED DESCRIPTION:
Pressure ulcers are defined as areas of localised damage to the skin, muscle or underlying tissue, caused by shear, friction or unrelieved pressure, usually over bony prominences. They are associated with many health conditions that cause prolonged bed rest, immobility, inactivity or poor sensation and can significantly contribute to morbidity and mortality, particularly in the aged population. International prevalence rates range widely from 4.6%- 83.6% due to methodological differences and classification systems. In Singapore, a study on the prevalence of pressure ulcers in 3 hospitals revealed a prevalence of 9% to 14%.

Pressure ulcers often fail to heal in a timely and orderly manner, resulting in a chronic non-healing wound. Many intrinsic and extrinsic factors have been identified that can disrupt the wound healing processes of haemostasis, inflammation, proliferation, angiogenesis and remodelling. One of the factors gaining more interest for its impact on wound healing processes is nutritional status.

Arginine is a semi-essential amino acid because even though the body normally makes enough of it, supplementation is sometimes needed during critical illness and severe trauma. There have been numerous research studies focusing on using arginine to enhance wound healing and pressure ulcer prevention. It is required for promotion of nitrogen balance, cell proliferation, T lymphocyte function and collagen accumulation. It also changes into nitric oxide, which is known for its vasodilatory and angiogenic properties.

Glutamine is conditionally essential amino acid because it can be manufactured in the body, but under extreme physical stress the demand for glutamine exceeds the body's ability to make it. Adequate amounts of glutamine are generally obtained through diet alone because the body is also able to make glutamine on its own. Certain medical conditions, including injuries, surgery, infections, and prolonged stress, can deplete glutamine levels. Since glutamine plays a key role in the immune system, a deficiency in this nutrient can significantly slow the healing process.

Beta-hydroxy-Beta methylbutyrate (HMB) is a metabolite of leucine, an essential amino acid. HMB supplementation was associated with increased muscle mass accretion. HMB appears to assert its effect via inhibiting muscle proteolysis and modulating protein turnover.

Recently, arginine has been found to accelerate wound healing in combination with HMB and glutamine. It was shown that healthy subjects who are supplemented orally with arginine had a significant rise in plasma arginine and ornithine levels that led to enhanced rate of collagen synthesis. In another recent study, a HMB/Arginine/Lysine mixture increased protein turnover in elderly patients over a year long period. However, there is no known randomised controlled trial done on patients with chronic hard to heal wounds in acute healthcare settings.

AIM To compare pressure ulcer healing rates in patients supplemented with a commercial HMB/Arginine/Lysine mixture (Abound) and standard high protein, high energy iso-nitrogenous medical nutritional supplements versus patients supplemented with only standard high protein, high energy iso-nitrogenous medical nutritional supplements.

OUTCOME INDICATORS

* Percentage change in wound size (length, depth, area)
* Percentage change in proportion of viable wound tissue (Refer to wound data collection for details)

The study will take on a comparative, randomised controlled trial design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pressure ulcers stage II, III or IV, non-healing admitted to Changi General Hospital for > 2 weeks
* Patients who are able to attend outpatient follow-up appointments for dietary and wound review

Exclusion Criteria:

* Age < 21 years old
* Poorly controlled Diabetic Patients (HbA1c >7.0%)
* Patients on Total Parenteral Nutrition
* Patients in MICU/ SICU/ Medically Unstable/ Palliative Care
* Patients with severe Sepsis
* Length of stay < 2 weeks
* Patients who require fluid restriction < 1L/d
* Patients on any other wound healing supplements (e.g. Zinc, Vitamin A and Vitamin C)
* Patients with lower extremity ulcers with untreated peripheral vascular disease
* Patients with deep tissue infection and/or requiring debridement of necrotic or sloughy tissue
* Patients unable to attend outpatient follow-up appointments
* Patients who cannot tolerate oral intake > 70% EER and/or Fluid intake 30ml/kg BW
* Patients who require protein restriction
* Patients who are unable to give consent (absence of next-of-kin)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvin Wong, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Baier S, Johannsen D, Abumrad N, Rathmacher JA, Nissen S, Flakoll P. Year-long changes in protein metabolism in elderly men and women supplemented with a nutrition cocktail of beta-hydroxy-beta-methylbutyrate (HMB), L-arginine, and L-lysine. JPEN J Parenter Enteral Nutr. 2009 Jan-Feb;33(1):71-82. doi: 10.1177/0148607108322403. PMID 19164608
- [Background] Smith HJ, Mukerji P, Tisdale MJ. Attenuation of proteasome-induced proteolysis in skeletal muscle by beta-hydroxy-beta-methylbutyrate in cancer-induced muscle loss. Cancer Res. 2005 Jan 1;65(1):277-83. PMID 15665304
- [Background] Eley HL, Russell ST, Baxter JH, Mukerji P, Tisdale MJ. Signaling pathways initiated by beta-hydroxy-beta-methylbutyrate to attenuate the depression of protein synthesis in skeletal muscle in response to cachectic stimuli. Am J Physiol Endocrinol Metab. 2007 Oct;293(4):E923-31. doi: 10.1152/ajpendo.00314.2007. Epub 2007 Jul 3. PMID 17609254
- [Background] Stechmiller JK, Childress B, Cowan L. Arginine supplementation and wound healing. Nutr Clin Pract. 2005 Feb;20(1):52-61. doi: 10.1177/011542650502000152. PMID 16207646
- [Background] Benati G, Delvecchio S, Cilla D, Pedone V. Impact on pressure ulcer healing of an arginine-enriched nutritional solution in patients with severe cognitive impairment. Arch Gerontol Geriatr Suppl. 2001;7:43-7. doi: 10.1016/s0167-4943(01)00120-0. No abstract available. PMID 11431045
- [Background] Desneves KJ, Todorovic BE, Cassar A, Crowe TC. Treatment with supplementary arginine, vitamin C and zinc in patients with pressure ulcers: a randomised controlled trial. Clin Nutr. 2005 Dec;24(6):979-87. doi: 10.1016/j.clnu.2005.06.011. Epub 2005 Nov 15. PMID 16297506
- [Derived] Wong A, Chew A, Wang CM, Ong L, Zhang SH, Young S. The use of a specialised amino acid mixture for pressure ulcers: a placebo-controlled trial. J Wound Care. 2014 May;23(5):259-60, 262-4, 266-9. doi: 10.12968/jowc.2014.23.5.259. PMID 24810310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 subjects were recruited between June 2010 to June 2011 and all subjects were inpatients of Changi General Hospital. 23 subjects completed the trial.
Pre-assignment Details: Subjects were randomly assigned to either arm after an initial assessment by PI and wound nurses. There is no wash out period for this trial
Groups:
- Abound: Active Arm : Abound x 2 sachets/d (Each sachet provides additional 7g L-Arginine, 7g L-Glutamine, 1.2 g HMB and 79 Kcal)
- Placebo: Placebo x 2 sachets/d
Period: Overall Study
Arm/Group | Abound | Placebo
Started | 12 | 14
Completed | 11 | 12
Not Completed | 1 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Abound; Placebo: Abound (7 g of Arginine, 7 g Glutamine and 1.2 g HMB) : Active Arm : Abound x 2 sachets/d (Each sachet provides additional 7g L-Arginine, 7g L-Glutamine, 1.2 g HMB and 79 Kcal) Placebo Arm: Abound(placebo) x 2 sachets/d
- Total: Total of all reporting groups
Arm/Group | Abound | Placebo | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 11 | 10 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 78.5 (18.4) | 74.3 (12.4) | 75.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 3 | 8 | 11
Region of Enrollment [Number; unit: participants]
  Singapore | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: % Viable Tissue
Description: -Percentage viable tissue after 2 weeks
  The estimated change in proportion of viable and non-viable tissue was determined using area derived from planimetry via acetate tracings. The description of viable tissue was taken to mean granulating (red) or epithelising (pink) tissue, and non-viable tissue were taken as necrotic (black) or sloughy (green or yellow) tissue.
Time Frame: weeks 1 to 2
Measure: Mean (Standard Error); unit: Percentage of viable tissue
Arm/Group | Abound | Placebo
Number analyzed (Participants) | 11 | 12
Percentage of viable tissue | 43.06 (8.43) | 25.94 (6.68)
Statistical Analysis 1: Comparison: Abound vs Placebo; Test type: Superiority or Other; p = 0.023, t-test, 2 sided

2. Primary Outcome: % Wound Area Week 1
Description: Percentage change in wound area after week 1
Time Frame: week 0 to 1
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Abound | Placebo
Number analyzed (Participants) | 11 | 12
percent change | -15.37 (7.64) | -13.68 (7.68)
Statistical Analysis 1: Comparison: Abound vs Placebo; Test type: Superiority or Other; p = 0.877, t-test, 2 sided

3. Primary Outcome: % Wound Area Week 2
Description: Percentage change in wound area after week 2
Time Frame: Weeks 1 to 2
Measure: Mean (Standard Error); unit: Percentage change
Arm/Group | Abound | Placebo
Number analyzed (Participants) | 11 | 12
Percentage change | -27.50 (10.11) | -37.54 (7.33)
Statistical Analysis 1: Comparison: Abound vs Placebo; Test type: Superiority or Other; p = 0.44, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Abound | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

LIMITATIONS AND CAVEATS:
Limitations of trial include small sample size and it was difficult to standardise wound care regimen as the pressure ulcers were of different stages and locations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes